CLINICAL TRIAL: NCT03310463
Title: Evaluation of the Pharmacokinetics, Safety, and Tolerability of Intravenous ETX2514 and Sulbactam Administered Concurrently to Subjects With Various Degrees of Renal Impairment and Healthy Matched Control Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS2514-2017-0002
Record Dates: First submitted 2017-09-25; First posted 2017-10-16 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Acinetobacter Baumannii Infection
Keywords: infection; gram-negative bacterium; renal impairment
MeSH Terms: conditions — Infections; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1, Normal Renal Function (Experimental): Healthy control participants matched to participants enrolled in Cohort 4 (creatinine clearance ≥90 milliliters per minute [mL/min] estimated by the Cockcroft-Gault equation) will receive ETX2514SUL as a single dose of up to 1000 milligrams (mg) ETX2514 and 1000 mg sulbactam given by concurrent 3-hour intravenous (IV) infusion.
  Interventions: Drug: ETX2514SUL
- Cohort 2, Mild Renal Impairment (Experimental): Participants with mild renal impairment (estimated glomerular filtration rate [eGFR] ≥60 to <90 mL/min/1.73 meters squared [m^2] calculated by the Modified Diet in Renal Disease [MDRD] equation) will receive ETX2514SUL as a single dose of up to 1000 mg ETX2514 and 1000 mg sulbactam given by concurrent 3-hour IV infusion.
  Interventions: Drug: ETX2514SUL
- Cohort 3, Moderate Renal Impairment (Experimental): Participants with moderate renal impairment (eGFR ≥30 to <60 mL/min/1.73 m^2 calculated by the MDRD equation) will receive ETX2514SUL as a single dose of up to 1000 mg ETX2514 and 1000 mg sulbactam given by concurrent 3-hour IV infusion.
  Interventions: Drug: ETX2514SUL
- Cohort 4, Severe Renal Impairment (Experimental): Participants with severe renal impairment (eGFR <30 mL/min/1.73 m^2 calculated by the MDRD equation) and not on hemodialysis (HD) will receive ETX2514SUL as a single dose of up to 1000 mg ETX2514 and 1000 mg sulbactam given by concurrent 3-hour IV infusion.
  Interventions: Drug: ETX2514SUL
- Cohort 5, ESRD on a Stable HD Regimen (Experimental): Participants with end-stage renal disease (ESRD) on a stable HD regimen (determined by medical history) will receive ETX2514SUL as a single dose of up to 1000 mg ETX2514 and 1000 mg sulbactam given by concurrent 3-hour IV infusion.
  Interventions: Drug: ETX2514SUL

INTERVENTIONS:
Drug: ETX2514SUL — Single dose of up to 1000 mg ETX2514 and 1000 mg sulbactam given by concurrent 3-hr IV infusion

SUMMARY:
This research project is being conducted to look at the pharmacokinetics (PK; how the human body processes a substance), safety, and tolerability of a single dose of ETX2514 and sulbactam (ETX2514SUL) when concurrently administered by separate intravenous (IV) infusion in participants with various degrees of renal impairment (RI), in participants with end-stage renal disease (ESRD) who are on hemodialysis (HD), and in healthy matched control participants with normal renal function.

DETAILED DESCRIPTION:
This Phase 1, open-label, non-randomized study evaluates the PK, safety, and tolerability of a single concurrent IV infusion of ETX2514SUL in participants with various degrees of RI, in participants with ESRD who are on HD, and in healthy matched control participants with normal renal function.

Participants will be enrolled into five cohorts, according to renal function status, and will receive an IV infusion of ETX2514SUL (single dose of up to 1000 milligrams [mg] ETX2514 and 1000 mg sulbactam given by concurrent 3-hour IV infusion). Participants in Cohort 5 will receive the ETX2514SUL infusion both post-HD (Period 1) and pre-HD (Period 2).

ELIGIBILITY:
Inclusion Criteria:

To qualify for enrollment in this study, each participant must meet the inclusion criteria for all participants, as well as all inclusion criteria specified for either healthy participants, participants with renal impairment (RI), or participants with end-stage renal disease (ESRD) requiring hemodialysis (HD):

All Participants (Cohorts 1-5)

* Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements and study-related procedures
* Willing to be confined to the Clinical Research Unit for the entire duration required by the protocol, able to comply with all study-related requirements and able to adhere to study restrictions and visit schedules
* Male or female, between 18 and 75 years of age (inclusive) at the time of Screening
* Body mass index (BMI) between 18 and 40 kilograms per meters squared (kg/m^2) (inclusive) at the time of Screening
* Female participants must:

  * be non-pregnant and non-lactating;
  * be either postmenopausal (defined as amenorrhea for ≥12 months with a confirmed follicle stimulating hormone [FSH] ≥40 milli International Units per milliliter [mIU/mL]), surgically sterile (defined as having undergone hysterectomy and/or bilateral oophorectomy), practice total abstinence from sexual intercourse as the preferred lifestyle (periodic abstinence is not acceptable), or agree to use an appropriate method of birth control consistently throughout the study and continue to use this method for 30 days (or 5 half-lives, whichever is longer) after study drug administration;
  * Hormonal contraception and double barrier methods of non-hormonal contraception are permitted in this study. Acceptable forms of contraception include the following:

    * oral, implantable, transdermal, injectable, or intravaginal hormonal contraception used consistently for at least 1 month prior to Screening;
    * intrauterine device;
    * female condom with spermicide (cream, spray, gel, suppository, contraceptive sponge, or polymer film);
    * contraceptive sponge with condom;
    * diaphragm with spermicide (with or without a condom);
    * cervical cap with spermicide (with or without a condom);
    * male sexual partner who agrees to use a male condom in addition to female participant's use of spermicide (cream, spray, gel, suppository, contraceptive sponge, or polymer film);
    * male sexual partner who has been vasectomized for at least 3 months prior to Screening and who has obtained a follow-up negative sperm count;
    * bilateral tubal ligation;
    * Essure® procedure.
* Male participants who are sexually active with a partner of child-bearing potential must either be sterile (vasectomy with history of a negative sperm count following the procedure); practice total abstinence from sexual intercourse as the preferred lifestyle (periodic abstinence is not acceptable); use a male condom with any sexual activity; or agree to use a birth control method considered to be appropriate by the Investigator (such as one of the methods identified above for female participants of childbearing potential) from the time of Screening until 90 days after study drug administration. Male participants must agree not to donate sperm for a period of 90 days after study drug administration.

Healthy Participants (Cohort 1)

In addition to the criteria specified above for all participants, healthy participants must also meet the following inclusion criteria:

* Considered by the Investigator to be healthy, based on medical and surgical history, and a complete physical examination including vital signs (VS), a 12-lead electrocardiogram (ECG), and laboratory test results. A single repeat assessment is permitted for any VS, ECG, or laboratory parameter required for enrollment.
* Estimated creatinine clearance ≥90 milliliters per minute (mL/min) (based on Cockcroft-Gault equation) determined at Screening
* Matched demographically with a participant in Cohort 4 (severe RI) according to gender, BMI (±20%), and age (±10 years)
* Has been a non-smoker (tobacco) for at least 30 days
* Healthy participants must not be taking any prescribed or non-prescribed medications, including vitamins and other dietary or herbal supplements, unless permitted (e.g., hormonal contraception, low dose aspirin [81 milligrams (mg)/day or less]).

Participants with RI (Cohorts 2-4)

In addition to the criteria specified above for all participants, participants with RI must also meet the following inclusion criteria:

* Participant has been diagnosed with RI in one of the three groups (e.g., mild, moderate, or severe) as defined by estimated glomerular filtration rate using the Modified Diet in Renal Disease equation at Screening
* Considered by the Investigator to be clinically stable with respect to underlying RI, based on medical evaluation that includes medical and surgical history, as well as a complete physical examination including VS, ECG, and laboratory test results. A single repeat assessment is permitted for any VS, ECG, or laboratory parameter required for enrollment.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin within 1.5 × upper limit of normal (ULN) at Screening
* Participants with renal impairment will be allowed to take their chronic medications unless excluded by the protocol. Excluded medications are restricted starting 7 days prior to study drug administration on Day 1 until the end of study visit. The occasional use of acetaminophen (≤2 grams per day) is permitted at the discretion of the Investigator.
* Will smoke ≤10 cigarettes (and consume no more than the cumulative equivalent amount of nicotine) per day from Screening until the Follow-up visit

Participants with ESRD Requiring HD (Cohort 5)

In addition to the criteria specified above for all participants, participants with ESRD requiring HD must also meet the following criteria:

* Diagnosed with ESRD and is on a stable HD regimen, defined as kt/V ≥1.2 within 3 months prior to Screening
* Typically attends 3 HD treatments per week within the 3 months prior to Screening, as determined by the Investigator
* Considered by the Investigator to be clinically stable with respect to underlying ESRD, based on medical evaluation that includes medical and surgical history, and a complete physical examination including VS, ECG, and laboratory test results. A single repeat assessment is permitted for any laboratory, ECG, or VS parameter required for enrollment.
* AST, ALT, and total bilirubin within 1.5 × ULN at Screening
* Participants with ESRD will be allowed to take their chronic medications unless excluded by the protocol. Excluded medications are restricted starting 7 days prior to study drug administration on Day 1 until the end of study visit. The occasional use of acetaminophen (≤2 grams per day) is permitted at the discretion of the Investigator.
* Will smoke ≤10 cigarettes (and consume no more than the cumulative equivalent amount of nicotine) per day from Screening until the Follow-up visit.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria for all participants, or any of the criteria specified for their respective renal function cohort, are not eligible for study enrollment.

All Participants (Cohorts 1-5)

* Known sensitivity or idiosyncratic reaction to any compound present in ETX2514 or sulbactam, its related compounds, or any compound listed as being present in the study formulation
* Participants with a history of hypersensitivity or serious adverse reaction to β-lactam agents (penicillin, cephalosporin, carbapenem, or sulbactam)
* Pregnant (positive pregnancy test) or lactating women at Screening or Day -1. If serum human chorionic gonadotropin (hCG) pregnancy test results are indeterminate, follow-up testing should be performed to determine eligibility.
* All female participants will not be pregnant and will have a negative pregnancy test at Screening and Day -1, with the following exception: females receiving dialysis with an indeterminate pregnancy test result or persistently low hCG resulting in a false positive pregnancy test may be included in the study at the discretion of the Investigator and notification of the Sponsor. Postmenopausal participants with a result outside the post-menopausal range or an indeterminate pregnancy test will undergo additional testing for FSH to confirm postmenopausal status prior to study enrollment.
* Any clinically significant (CS) concomitant disease or condition (including treatment for such conditions) that, in the opinion of the Investigator, could either interfere with the study drug or pose an unacceptable risk to the participant
* Any other CS abnormalities in laboratory test results at Screening that would, in the opinion of the Investigator, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
* Uncontrolled medical condition (treated or untreated) considered to be CS by the Investigator
* Treatment with another investigational drug or device study within 30 days (or 5 half-lives, whichever is longer) prior to study drug administration on Day 1
* Participant has taken probenecid within 30 days prior to study drug administration on Day 1
* Has experienced an illness that is considered by the Investigator to be CS within 2 weeks of study drug administration on Day 1
* Has donated or lost a significant volume (>450 mL) of blood within 56 days or plasma within 7 days prior to Day -1
* Participated in strenuous exercise from 48 hours prior to Day -1 or during the study through the final end of study assessment
* Exclusion criteria for ECG at Screening, Day -1, and Day 1 predose (a single repeat is allowed for eligibility determination, with Investigator discretion for RI and ESRD participants):

  * Evidence of previous myocardial infarction (did not include ST segment changes associated with repolarization)
  * Any conduction abnormality (including but not specific to atrioventricular block [2nd degree or higher], Wolff Parkinson White syndrome [unless curative radio ablation therapy])
  * Sinus pauses >3 seconds
  * Any significant arrhythmia or conduction abnormality, which, in the opinion of the Investigators and Medical Monitor (MM), interfered with the safety for the individual participant
  * Non-sustained or sustained ventricular tachycardia (≥3 consecutive ventricular ectopic beats)
* Any other reason that would render the participant unsuitable for study enrollment at the discretion of the Investigator

Healthy Participants (Cohort 1)

Healthy participants will be excluded from the study if they meet any of the following criteria:

* The participant's systolic blood pressure was outside the range of 90 to 150 millimeters per mercury (mmHg), diastolic blood pressure was outside the range of 40 to 95 mmHg or heart rate was outside the range of 45 to 100 beats per minute at Screening.
* Positive test for drugs of abuse and/or positive alcohol test
* Positive test at Screening for any of the following: Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV), or human immunodeficiency virus (HIV)

Participants with RI (Cohorts 2-4)

Participants with RI will be excluded from the study if they meet any of the following criteria:

* Positive test for drugs of abuse and/or positive alcohol test if not accounted for by a prescription medication. Participants with a positive test based on a prescribed medication may be enrolled.
* Acute exacerbation of RI or unstable renal function, as determined by the Investigator, from Screening to Day 1
* Hemoglobin concentration <9.0 grams per deciliter (g/dL) at Screening
* Cohorts 2-4: Positive test at Screening for HBsAg or HIV
* Cohorts 2 and 3: Positive test at Screening for HCV. If a participant with severe RI (Cohort 4) has positive test results for HCV but liver function tests are otherwise not CS, the participant may be included at the Investigator's discretion (this provision does not apply to participants with mild or moderate RI [Cohorts 2 or 3]).

Participants with ESRD Requiring HD (Cohort 5)

Participants with ESRD will be excluded from the study if they meet any of the following criteria:

* Positive test for drugs of abuse and/or positive alcohol test if not accounted for by a prescription medication. Participants with a positive test based on a prescribed medication may be enrolled.
* Hemoglobin concentration <9.0 g/dL at Screening
* Positive test at Screening for HBsAg or HIV. If a participant with ESRD has positive test results for HCV but liver function tests are otherwise not clinically significant, the participant may be included at the Investigator's discretion.
* Receiving blood purification therapy other than HD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Mean maximum observed drug concentration (Cmax) in blood: Cohorts 1 and 2 | Days 1 to 3: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose")
  Venous blood will be collected for ETX2514SUL pharmacokinetic (PK) analyses.
Mean Cmax in blood: Cohorts 3 and 4 | Days 1 to 4: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose")
  Venous blood will be collected for ETX2514SUL PK analyses.
Mean Cmax in blood: Cohort 5 | Days 1 to 4. Period 1 (post-hemodialysis): predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Period 2 (pre-hemodialysis): approximately 4, 5, 6, and 7 hours after the start of infusion
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines. Hemodialysis will be started approximately 1 hour after the end of infusion. If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session.
Mean time to reach the maximum concentration (tmax) in blood: Cohorts 1 and 2 | Days 1 to 3: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose")
  Venous blood will be collected for ETX2514SUL PK analyses.
Mean tmax in blood: Cohorts 3 and 4 | Days 1 to 4: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose")
  Venous blood will be collected for ETX2514SUL PK analyses.
Mean tmax in blood: Cohort 5 | Days 1 to 4. Period 1 (post-hemodialysis): predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Period 2 (pre-hemodialysis): approximately 4, 5, 6, and 7 hours after the start of infusion
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines. Hemodialysis will be started approximately 1 hour after the end of infusion. If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session.
Mean AUC0-24 in blood: Cohorts 1 and 2 | Days 1 to 3: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose")
  AUC0-24 is defined as the area under the concentration versus time curve from time zero to 24 hours postdose. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-48 in blood: Cohorts 1 and 2 | Days 1 to 3: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose")
  AUC0-48 is defined as the area under the concentration versus time curve from time zero to 48 hours postdose. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-last in blood: Cohorts 1 and 2 | Days 1 to 3: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose")
  AUC0-last is defined as the area under the concentration versus time curve from time zero to the time of the last quantifiable concentration after dosing. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-∞ in blood: Cohorts 1 and 2 | Days 1 to 3: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose")
  AUC0-∞ is defined as the area under the concentration versus time curve from time zero extrapolated to infinity. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-24 in blood: Cohorts 3 and 4 | Days 1 to 4: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose")
  AUC0-24 is defined as the area under the concentration versus time curve from time zero to 24 hours postdose. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-48 in blood: Cohorts 3 and 4 | Days 1 to 4: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose")
  AUC0-48 is defined as the area under the concentration versus time curve from time zero to 48 hours postdose. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-60 in blood: Cohorts 3 and 4 | Days 1 to 4: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose")
  AUC0-60 is defined as the area under the concentration versus time curve from time zero to 60 hours. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-last in blood: Cohorts 3 and 4 | Days 1 to 4: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose")
  AUC0-last is defined as the area under the concentration versus time curve from time zero to the time of the last quantifiable concentration after dosing. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-∞ in blood: Cohorts 3 and 4 | Days 1 to 4: predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose")
  AUC0-∞ is defined as the area under the concentration versus time curve from time zero extrapolated to infinity. Venous blood will be collected for ETX2514SUL PK analyses.
Mean AUC0-24 in blood: Cohort 5 | Days 1 to 4. Periods 1 (post-hemodialysis): predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Period 2 (pre-hemodialysis): approximately 4, 5, 6, and 7 hours after the start of infusion
  AUC0-24 is defined as the area under the concentration versus time curve from time zero to 24 hours postdose. Venous blood will be collected for ETX2514SUL PK analyses in Period 1. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines. Hemodialysis will be started approximately 1 hour after the end of infusion. If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session.
Mean AUC0-48 in blood: Cohort 5 | Days 1 to 4. Periods 1 (post-hemodialysis): predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Period 2 (pre-hemodialysis): approximately 4, 5, 6, and 7 hours after the start of infusion
  AUC0-48 is defined as the area under the concentration versus time curve from time zero to 48 hours postdose. Venous blood will be collected for ETX2514SUL PK analyses in Period 1. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines. Hemodialysis will be started approximately 1 hour after the end of infusion. If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session.
Mean AUC0-60 in blood: Cohort 5 | Days 1 to 4. Periods 1 (post-hemodialysis): predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Period 2 (pre-hemodialysis): approximately 4, 5, 6, and 7 hours after the start of infusion
  AUC0-60 is defined as the area under the concentration versus time curve from time zero to 60 hours postdose. Venous blood will be collected for ETX2514SUL PK analyses in Period 1. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines. Hemodialysis will be started approximately 1 hour after the end of infusion. If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session.
Mean AUC0-last in blood: Cohort 5 | Days 1 to 4. Periods 1 (post-hemodialysis): predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Period 2 (pre-hemodialysis): approximately 4, 5, 6, and 7 hours after the start of infusion
  AUC0-last is defined as the area under the concentration versus time curve from time zero to the time of the last quantifiable concentration after dosing. Venous blood will be collected for ETX2514SUL PK analyses in Period 1. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines. Hemodialysis will be started approximately 1 hour after the end of infusion. If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session.
Mean AUC0-∞ in blood: Cohort 5 | Days 1 to 4. Periods 1 (post-hemodialysis): predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Period 2 (pre-hemodialysis): approximately 4, 5, 6, and 7 hours after the start of infusion
  AUC0-∞ is defined as the area under the concentration versus time curve from time zero extrapolated to infinity. Venous blood will be collected for ETX2514SUL PK analyses in Period 1. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous. Hemodialysis will be started approximately 1 hour after the end of infusion. If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session.
Mean terminal elimination rate constant (λz) in blood: Cohorts 1 and 2 | Days 1 to 3
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 48 hours post infusion could fall on Day 3.
Mean λz in blood: Cohorts 3 and 4 | Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean λz in blood: Cohort 5 | Periods 1 (post-hemodialysis) and 2 (pre-hemodialysis): Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1 at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines at approximately 4, 5, 6, and 7 hours after the start of infusion (where hemodialysis will be started approximately 1 hour after the end of infusion). If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean terminal half life (t1/2) in blood: Cohorts 1 and 2 | Days 1 to 3
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 48 hours post infusion could fall on Day 3.
Mean t1/2 in blood: Cohorts 3 and 4 | Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean t1/2 in blood: Cohort 5 | Periods 1 (post-hemodialysis) and 2 (pre-hemodialysis): Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1 at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines at approximately 4, 5, 6, and 7 hours after the start of infusion (where hemodialysis will be started approximately 1 hour after the end of infusion). If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean total clearance (CL) from blood: Cohorts 1 and 2 | Days 1 to 3
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 48 hours post infusion could fall on Day 3.
Mean CL from blood: Cohorts 3 and 4 | Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean CL in blood: Cohort 5 | Periods 1 (post-hemodialysis) and 2 (pre-hemodialysis): Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1 at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines at approximately 4, 5, 6, and 7 hours after the start of infusion (where hemodialysis will be started approximately 1 hour after the end of infusion). If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean volume of distribution in the terminal elimination phase (Vz) in blood: Cohorts 1 and 2 | Days 1 to 3
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, and 48 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 48 hours post infusion could fall on Day 3.
Mean Vz in blood: Cohorts 3 and 4 | Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, and 60 hours after the start of infusion ("postdose"). Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean Vz in blood: Cohort 5 | Periods 1 (post-hemodialysis) and 2 (pre-hemodialysis): Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1 at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines at approximately 4, 5, 6, and 7 hours after the start of infusion (where hemodialysis will be started approximately 1 hour after the end of infusion). If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean cumulative amount of drug excreted in urine (Aeu): Cohorts 1 and 2 | Days 1 and 2
  Urine for ETX2514SUL PK analyses will be collected continuously from participants capable of producing urine at the following intervals: predose (a single void within 30 minutes prior to the start of infusion) and 0 to 4, 4 to 8, 8 to 12, and 12 to 24 hours after the start of infusion. Infusion can begin at any time on Day 1; thus, 24 hours post infusion could fall on Day 2.
Mean Aeu: Cohorts 3 and 4 | Days 1 to 4
  Urine for ETX2514SUL PK analyses will be collected continuously from participants capable of producing urine at the following intervals: predose (a single void within 30 minutes prior to the start of infusion), and 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 60 hours after the start of infusion. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean renal clearance (CLR): Cohorts 1 and 2 | Days 1 and 2
  Urine for ETX2514SUL PK analyses will be collected continuously from participants capable of producing urine at the following intervals: predose (a single void within 30 minutes prior to the start of infusion) and 0 to 4, 4 to 8, 8 to 12, and 12 to 24 hours after the start of infusion. Infusion can begin at any time on Day 1; thus, 24 hours post infusion could fall on Day 2.
Mean CLR: Cohorts 3 and 4 | Days 1 to 4
  Urine for ETX2514SUL PK analyses will be collected continuously from participants capable of producing urine at the following intervals: predose (a single void within 30 minutes prior to the start of infusion), and 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 60 hours after the start of infusion. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean fraction of the dose renally eliminated (Feu): Cohorts 1 and 2 | Days 1 and 2
  Urine for ETX2514SUL PK analyses will be collected continuously from participants capable of producing urine at the following intervals: predose (a single void within 30 minutes prior to the start of infusion) and 0 to 4, 4 to 8, 8 to 12, and 12 to 24 hours after the start of infusion. Infusion can begin at any time on Day 1; thus, 24 hours post infusion could fall on Day 2.
Mean Feu: Cohorts 3 and 4 | Days 1 to 4
  Urine for ETX2514SUL PK analyses will be collected continuously from participants capable of producing urine at the following intervals: predose (a single void within 30 minutes prior to the start of infusion), and 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 60 hours after the start of infusion. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean amount dialyzed (AHD): Cohort 5 | Periods 1 (post-hemodialysis) and 2 (pre-hemodialysis): Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1 at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines at approximately 4, 5, 6, and 7 hours after the start of infusion (where hemodialysis will be started approximately 1 hour after the end of infusion). If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Mean fraction of the dose removed by hemodialysis (FHD): Cohort 5 | Periods 1 (post-hemodialysis) and 2 (pre-hemodialysis): Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1 at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines at approximately 4, 5, 6, and 7 hours after the start of infusion (where hemodialysis will be started approximately 1 hour after the end of infusion). If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.
Estimated hemodialysis (HD) recovery clearance (CLD Recovery): Cohort 5 | Periods 1 (post-hemodialysis) and 2 (pre-hemodialysis): Days 1 to 4
  Venous blood will be collected for ETX2514SUL PK analyses in Period 1 at predose, and 0.5, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 60 hours after the start of infusion. Blood will be collected for ETX2514SUL PK analyses in Period 2 from arterial and venous lines at approximately 4, 5, 6, and 7 hours after the start of infusion (where hemodialysis will be started approximately 1 hour after the end of infusion). If the hemodialysis session takes longer than 7 hours after the start of infusion, a final sample will be collected at the end of the hemodialysis session. Infusion can begin at any time on Day 1; thus, 60 hours post infusion could fall on Day 4.

SECONDARY OUTCOMES:
Number of participants with any non-serious adverse event (AE) | Cohorts 1 and 2: Days 1, 2, 3, and 7. Cohorts 3 and 4: Days 1, 2, 3, 4, and 7. Cohort 5: Period 1: Days 1, 2, 3, and 4; Washout. Period 2: Days -1, 2, 3, 4, and 7
  An AE is defined as any untoward medical occurrence in a participant enrolled into this study regardless of its causal relationship to study drug.
Number of participants with any serious adverse event (SAE) | Cohorts 1 and 2: Days 1, 2, 3, and 7. Cohorts 3 and 4: Days 1, 2, 3, 4, and 7. Cohort 5: Period 1: Days 1, 2, 3, and 4; Washout. Period 2: Days -1, 2, 3, 4, and 7.
  An SAE is defined as any event that results in death; is immediately life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
Number of participants with an adverse event of the indicated causality and severity | Cohorts 1 and 2: Days 1, 2, 3, and 7. Cohorts 3 and 4: Days 1, 2, 3, 4, and 7. Cohort 5: Period 1: Days 1, 2, 3, and 4; Washout. Period 2: Days -1, 2, 3, 4, and 7
  An AE is defined as any untoward medical occurrence in a participant enrolled into this study regardless of its causal relationship to study drug. Wherever possible, the severity of all AEs will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03). The Investigator's assessment of causality must be provided for all AEs. The causality is the determination of whether there exists a reasonable possibility that the study drug itself caused or contributed to an AE.
Number of participants with abnormal, clinically significant physical examination findings at the indicated time points | Cohorts 1 and 2: Screening; Days -1 and 7. Cohorts 3 and 4: Screening; Days -1 and 7. Cohort 5: Period 1: Screening; Day -1. Period 2: Day 7
  Clinical significance will be determined by the Investigator.
Number of participants with abnormal, clinically significant vital sign values at the indicated time points | Cohorts 1 and 2: Screening; Days -1, 1, 2, 3, and 7. Cohorts 3 and 4: Screening; Days -1, 1, 2, 3, 4, and 7. Cohort 5: Period 1: Screening; Days -1, 1, 2, 3, and 4. Period 2: Days -1, 1, 2, 3, 4, and 7.
  Clinical significance will be determined by the Investigator.
Change from Baseline in electrocardiogram (ECG) parameters at the indicated time points | Cohorts 1 and 2: Screening; Days -1, 1, and 7. Cohorts 3 and 4: Screening; Days -1, 1, and 7. Cohort 5: Period 1: Screening; Days -1 and 1. Period 2: Days -1, 1, and 7
  Change from Baseline is calculated as the post-Baseline value minus the Baseline value.
Number of participants with abnormal, clinically significant hematology and clinical chemistry laboratory values at the indicated time points | Cohorts 1 and 2: Screening; Days -1, 2, and 7. Cohorts 3 and 4: Screening; Days -1, 2, and 7. Cohort 5: Period 1: Screening; Days -1 and 2. Period 2: Days -1, 2, and 7
  Clinical significance will be determined by the Investigator.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - DaVita Clinical Research, Lakewood, Colorado
  - University of Miami, Division of Clinical Pharmacology, Miami, Florida
  - Davita Clinical Research, Minneapolis, Minnesota